CLINICAL TRIAL: NCT02091557
Title: CA 125 and VAS Pain Score Changes Following GnRH-analog Administration as ex Adiuvantibus Criteria to Diagnose Endometriosis as Cause of Chronic Pelvic Pain.
Brief Title: CA 125 and VAS Pain Score Changes to Diagnose Endometriosis
Status: Completed | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Other Study IDs: CA125_VAS_changes
Record Dates: First submitted 2014-03-15; First posted 2014-03-19 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Pelvic Pain; Endometriosis
Keywords: GnRH-a; endometriosis; chronic pelvic pain; VAS score; diagnostic accuracy
MeSH Terms: conditions — Pelvic Pain; Endometriosis | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GnRH-analogue: CA125 levels and VAS pain score changes will be assessed after GnRH-a administration in all patients
  Interventions: Drug: GnRH-analogue

INTERVENTIONS:
Drug: GnRH-analogue
  Other Names: LAD

SUMMARY:
To assess the diagnostic accuracy for the noninvasive detection of pelvic endometriosis of the combination of two simple parameters: modifications of serum CA 125 and VAS pain score following one dose of GnRH-analog (GnRH-a).

DETAILED DESCRIPTION:
Between January 2010 and January 2014, women scheduled for a diagnostic laparoscopy for CPP at our Department will be enrolled in the current prospective observational study. For these patients, laparoscopy represents the last diagnostic step after medical history negative for gastrointestinal, urological, musculoskeletal and psychoneurological disorders related to pelvic pain, physical examination, ultrasonographic assessment and laboratory testing. From all patients, at enrollment, blood samples for serum CA125 determination will be taken during the early follicular phase (2nd-3rd day of the menstrual cycle) and VAS score for menstrual pain will be assessed. Electrochemiluminescence immunoassay (Immunoassay Elecsys Systems, Roche Diagnostics, Italy) for serum CA125 assay will be used (kit coefficient of variation between-run 0.0% and within-run 2.0%).

During the time passed on surgery waiting list, patients will received leuprolide acetate depot (LAD) at a dose of 3.75 mg IM at the 21st day of the menstrual cycle. One month later LAD administration, serum CA125 levels and VAS score will be assessed again, and then the surgical procedure will be performed in all these patients.

After laparoscopy and definitive histological examination, the population initially enrolled will be sub-grouped according to endometriosis diagnosis in two groups, i.e. group 1 (subjects with endometriosis) and group 2 (subjects without endometriosis).

ELIGIBILITY:
Inclusion Criteria:

* chronic pelvic pain

Exclusion Criteria:

* age less than 18 and greater than 38
* oligo-amenorrhea
* use of hormone medications (including oral contraceptives pill, progestogens, and so on)
* conditions affecting serum CA125 levels (such as, pregnancy, ovarian endometrioma seen at ultrasonography, pelvic inflammatory diseases, neoplasm, tuberculosis, hepatitis, peritonitis, recent abdominal surgery and pelvic organic disease)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic pelvic pain
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of composite measure (serum CA 125 levels and VAS pain score changes following one dose of GnRH-a) | One month after LAD administration
  Diagnostic accuracy (specificity, sensitivity, AUC and cut off levels) of the modifications of serum CA 125 levels and VAS pain score following one dose of LAD (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy

REFERENCES:
- [Background] Venturella R., et al. CA 125 modifications throughout menstrual cycle and following GnRH-analog administration to diagnose endometriosis as cause of chronic pelvic pain.A prospective controlled study. Journal of Endometriosis 2011; 3(3): 151 - 158. DOI: 10.5301/JE.2011.8911